CLINICAL TRIAL: NCT02429609
Title: Exploring the Psychophysics of Keratoconus Using the Moorfields Acuity Chart
Acronym: MACK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Moorfields Eye Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ANDO1009
Record Dates: First submitted 2015-04-09; First posted 2015-04-29 (Estimated); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Keratoconic Subjects

STUDY DESIGN:
Intervention Model Description: This in a basic science exploratory study to examine the effect of keratoconus on visual acuity as measured using pseudo-high-pass filtered optotypes. The MAC will be compared with the standard charts currently used to monitor visual acuity (logMAR chart) and contrast sensitivity (Pelli-Robson). "Researcher effects" and "researcher bias" will be controlled by setting a written protocol for all testing procedures. Each procedure will be standardised and random checks will be made by the chief investigator on all anonymous record sheets. Neither the chief investigator nor the co-researchers will act as participants for this study.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Keratoconic subjects (Experimental): 1. Short clinical interview (Questions pertaining to ocular and systemic health, medications, family history and date of birth). (approx. 2 minutes)
  2. Visual acuity measurement using EDTRS chart at 4 m (approx. 4 minutes)
  3. Refraction: retinoscopy and subjective, at 4m (approx. 10 minutes)
  4. Anterior eye examination (approx. 4 minutes)
  5. Fundus examination using binocular indirect ophthalmoscopy or a standard ophthalmoscope - to screen for eye disease that is likely to affect visual ability in this study. (approx. 5 minutes)
  6. Corneal topography measurement with an Oculus Pentacam (Oculus Gmbh., Germany). (approx. 5 minutes)
  Two measurements of visual acuity will be made:
  1. Standard ETDRS logMAR acuity measurement (5 minutes)
  2. Vanishing Optotype logMAR acuity measurement (5 minutes)
  Interventions: Device: Moorfields Acuity Chart
- Healthy subjects (Experimental): 1. Short clinical interview (Questions pertaining to ocular and systemic health, medications, family history and date of birth). (approx. 2 minutes)
  2. Visual acuity measurement using EDTRS chart at 4 m (approx. 4 minutes)
  3. Refraction: retinoscopy and subjective, at 4m (approx. 10 minutes)
  4. Anterior eye examination (approx. 4 minutes)
  5. Fundus examination using binocular indirect ophthalmoscopy or a standard ophthalmoscope - to screen for eye disease that is likely to affect visual ability in this study. (approx. 5 minutes)
  6. Corneal topography measurement with an Oculus Pentacam (Oculus Gmbh., Germany). (approx. 5 minutes)
  Two measurements of visual acuity will be made:
  1. Standard ETDRS logMAR acuity measurement (5 minutes)
  2. Vanishing Optotype logMAR acuity measurement (5 minutes)
  Interventions: Device: Moorfields Acuity Chart

INTERVENTIONS:
Device: Moorfields Acuity Chart

SUMMARY:
The measurement of visual acuity is made using black letters of varying size superimposed on a uniform white background. The objective is to determine the smallest letter, or optotype, that can be correctly identified. One limitation of current tests is the variability of measurements, this making it difficult for clinicians to determine if changes in visual acuity are related to ocular disease. This variability has been attributed to the design of current optotypes, in particular their differing legibilities. Our group has recently demonstrated that a new type of letter chart (Moorfields Acuity Chart), containing letters with a black core and a white border presented on a grey background, reduces the variability of visual acuity measurements. In this study the investigators wish to determine if changes in vision owing to keratoconus, a disease that causes the cornea to adopt an irregular shape, may be detected more easily using the Moorfields Acuity Chart compared with conventional letter charts.

ELIGIBILITY:
Keratoconic subjects (50):

* Age 18-40 years.
* The presence of keratoconus in at least one eye.
* The absence of significant media opacities (e.g. cataract, corneal scarring).
* The absence of any other ocular pathology (e.g. glaucoma, diabetic retinopathy, uveitis).
* The absence of amblyopia in the test eye.
* No previous ocular surgery (e.g. corneal crosslinking, cataract surgery, etc.)
* Best corrected visual acuity better than or equal to 6/60 (1.0 logMAR).
* Pupil diameter ≥3 mm and ≤7 mm in normal room illumination.

Healthy subjects (30):

* Age 18-35 years.
* The absence of clinically significant keratoconus.
* The absence of significant media opacities. (e.g. cataract, corneal scarring).
* The absence of any other ocular pathology (e.g. glaucoma, diabetic retinopathy, uveitis).
* The absence of amblyopia in the test eye.
* No previous ocular surgery (e.g. corneal crosslinking, cataract surgery, etc.)
* Best corrected visual acuity better than or equal to 6/9 (0.1 logMAR).
* Pupil diameter ≥3 mm and ≤7 mm in normal room illumination.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2015-04-15 (Actual); Primary Completion 2016-04-30 (Actual); Study Completion 2016-04-30 (Actual)

PRIMARY OUTCOMES:
The relative difference in visual acuity measurement between subjects with and without keratoconus when examined with different types of visual acuity chart. | 9 months

SECONDARY OUTCOMES:
The relationship (if any) between optical imperfections (high order aberrations) and measurements of visual acuity when measured using different test chart designs. | 9 months